CLINICAL TRIAL: NCT04041102
Title: Natural History Study of Infantile and Juvenile GM1 Gangliosidosis (GM1) Patients
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Passage Bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ODC-NHS-GM1-001-01
Record Dates: First submitted 2019-07-16; First posted 2019-08-01 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: GM1 Gangliosidosis
Keywords: GM1; GM1 gangliosidosis; GM1 Type 1; GM1 Type 2; GM1 gangliosidosis Type 1; GM1 gangliosidosis Type 2; GM1 natural history study; GM1 gangliosidosis natural history study; Lysosomal Storage Disorders; Lysosomal Disorders
MeSH Terms: conditions — Gangliosidosis, GM1; Lysosomal Storage Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The protocol includes the collection and biobank storage of several biofluid samples for future research. The samples include plasma/serum, cerebrospinal fluid (CSF; optional) and urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infantile (Type 1) or Juvenile (Type 2) GM1 Gangliosidosis: This study observes one cohort: up to 40 Infantile GM1 (Type 1) or Juvenile GM1 (Type 2) subjects.

SUMMARY:
Owing to the rarity, severity, speed of progression and fatal prognosis of infantile and juvenile GM1, there is a limited understanding of overall disease progression and meaningful outcome measures. This study aims to build a natural history data set through collection of a number of clinical, imaging, and laboratory assessments that may be specific predictors of GM1 disease progression and clinical outcome. Having a GM1 natural history data set can inform potential efficacy endpoints and biomarkers for future clinical trials.

This natural history study will follow up to 40 subjects diagnosed with GM1 gangliosidosis (up to 20 infantile (Type 1) and 20 late infantile/juvenile (Type 2)) for up to 3 years. Visits will be conducted every 6 months, during which several procedures will be performed and the data recorded in order to learn about the natural course of the disease, including changes in clinical and neurological assessments and electrophysiologic, imaging and biofluid biomarkers. Study procedures include: physical & neurological exam, blood & urine sample collection, questionnaires & assessments of development, seizure diary, ECHO, ECG, x-ray and ultrasound (if MRI not performed), EEG and genetic testing (if not already done).

The following procedures are subject to local/institutional policies and the medical discretion of the Study Physician: MRI, lumbar puncture (spinal tap) and General anesthesia/sedation (for MRI and LP).

ELIGIBILITY:
Inclusion Criteria:

1. Documentation/ Confirmation of reduced beta-galactosidase enzyme activity in leukocytes
2. Confirmed diagnosis of infantile or juvenile GM1 gangliosidosis with documentation of GLB1 mutations
3. Parent/Caregiver capable of providing informed consent (if cognitively able, child to provide assent as well)
4. Infantile (Type 1) GM1 subjects: Documented symptom onset by 6 months of age with significant hypotonia on exam or history elicited from parent(s)/ caregiver(s)
5. Juvenile (Type 2) GM1 subjects: Documented symptom onset after 6 months of age OR documented symptom onset prior to 6 months of age without significant hypotonia on exam or elicited from parent(s)/ caregiver(s)

Exclusion Criteria:

1. Enrollment in any other clinical study with an investigational product/ therapy (patients receiving miglustat off-label will be eligible)
2. Any clinically significant neurocognitive deficit not attributable to GM1 gangliosidosis or a secondary cause that may, in the opinion of the investigator, confound interpretation of study results
3. Any condition that, in the opinion of the investigator, would put the subject at undue risk or make it unsafe for the subject to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with a diagnosis of infantile (Type 1) or juvenile (Type 2) GM1 gangliosidosis.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Survival (Infantile GM1 population) | Baseline through 36 months (3 years)
  Survival will be evaluated at the baseline visit and each subsequent visit for 3 years. This outcome measure is considered a primary outcome measure for the infantile (Type 1) GM1 population and a secondary outcome measure for the juvenile (Type 2) GM1 population.
Presence of and dependence on feeding tube (Infantile GM1 population) | Baseline through 36 months (3 years)
  The presence of a feeding tube and dependence on the feeding tube, if applicable, will be evaluated at the baseline visit and each subsequent visit for 3 years. This outcome measure is considered a primary outcome measure for the infantile (Type 1) GM1 population and a secondary outcome measure for the juvenile (Type 2) GM1 population.
Change from baseline in standard scores for each domain on the Vineland-II (Juvenile GM1 population) | Baseline through 36 months (3 years)
  The Vineland Adaptive Behavior Scales, Second Edition (Vineland-II) is a standard assessment for measuring personal and social skills for children and adults (birth through 90 years of age). This assessment aids in diagnosis of intellectual and developmental disabilities or delays associated with a variety of diseases/disorders. The assessment includes 5 domains. Scores for each domain and a composite adaptive behavior score are then converted to standard scores with a range of 20 to 140, with a score of 140 correlating to a high adaptive level.
Change from baseline in total score for each sub-domain of the BSID-III OR the KABC-II (Juvenile GM1 population) | Baseline through 36 months (3 years)
  Based on the outcome of the Vineland-II, each subject will be given a developmental age score that will determine whether the Bayley Scale of Infant and Toddler Development, Third Edition (BSID-III) or the Kaufman Assessment Battery for Children, Second Edition (KABC-II) is administered. Children with a developmental age of 42 months or less will be administered the BSID-III and those with a developmental age of greater than 42 months will be administered the KABC-II.
  The BSID-III assesses 5 major areas of development. Each domain results in a raw score that is converted to a composite score. A higher composite score generally corresponds with higher function.
  The KABC-II assesses 4 major areas of intelligence and achievement in young children. Each domain results in a raw score that is converted to a standard score. Scores from 90-109 are generally considered average, with scores higher than 109 considered to be above average.

SECONDARY OUTCOMES:
Survival (Juvenile GM1 population) | Baseline through 36 months (3 years)
  Survival will be evaluated at the baseline visit and each subsequent visit for 3 years. This outcome measure is considered a primary outcome measure for the infantile (Type 1) GM1 population and a secondary outcome measure for the juvenile (Type 2) GM1 population.
Presence of and dependence on feeding tube (Juvenile GM1 population) | Baseline through 36 months (3 years)
  The presence of a feeding tube and dependence on the feeding tube, if applicable, will be evaluated at the baseline visit and each subsequent visit for 3 years. This outcome measure is considered a primary outcome measure for the infantile (Type 1) GM1 population and a secondary outcome measure for the juvenile (Type 2) GM1 population.
Change from baseline in total score for each sub-domain of the BSID-III OR the KABC-II (Infantile GM1 population) | Baseline through 36 months (3 years)
  See these outcome measures described above for full details.
  The BSID-III or the KABC-II will be evaluated at the baseline visit and each subsequent visit for 3 years. This outcome measure is considered a primary outcome measure for the juvenile (Type 2) GM1 population and a secondary outcome measure for the infantile (Type 1) GM1 population.
Change from baseline in the PedsQL total score | Baseline through 36 months (3 years)
  The Pediatric Quality of Life Inventory, Version 4.0 (PedsQL) is a 21 to 45-item assessment of quality of life over the previous 30 days, based on parent/caregiver report. The inventory consists of assessments for infants, toddlers, young children, children, teens and young adults, based on the age of the subject. A lower total score indicates higher quality of life.
Change from baseline in attainment and/or retention of six World Health Organization motor development milestones | Baseline through 36 months (3 years)
  Motor development will be assessed in terms of six developmental milestones: sitting without support, standing with assistance, hands-and-knee crawling, walking with assistance, standing alone, and walking alone. Each milestone will be assessed as either "achieved", "not achieved" or "achieved but lost" based on clinician observation as well as parent report.
Onset of and/or change in seizure activity over time | Baseline through 36 months (3 years)
  The change from baseline in presence/absence of seizures and frequency of seizures (if applicable) will be examined through review of seizure diaries recorded by parents over a three year period.
Change from baseline ECG | Baseline through 36 months (3 years)
  An electrocardiogram (ECG) is a test using electrodes attached to the subject's chest, arms, and legs to record the electrical activity in the heart and detect abnormalities. The clinician will note whether each ECG is normal or abnormal, and the results will be compared to the baseline ECG and tracked over time.
Change from baseline in bony structures of the spine using X-ray | Baseline through 36 months (3 years)
  A lateral spine plain film involves taking an X-ray of the subject's spine to determine if there are structural abnormalities. An X-ray of the spine will be performed at the baseline visit, then every 6 months for up to three years in order to assess changes.
Change from baseline in ECHO parameters over time | Baseline through 36 months (3 years)
  An echocardiogram (ECHO) uses ultrasound to produce images of the subject's heart. The ECHO report will be evaluated for changes from baseline through the course of the study.
Change from baseline EEG | Baseline through 36 months (3 years)
  An electroencephalogram (EEG) is a test using electrodes attached to the subject's scalp to detect abnormal activity in the brain. The EEG should be performed, if consent if provided, at each visit. The clinician will note whether each ECG is normal or abnormal, and the results will be compared to the baseline ECG and tracked over time.
Change from baseline in brain volume and volume of substructures measured using MRI | Baseline through 36 months (3 years)
  If consent if provided, magnetic resonance imaging (MRI) of the brain will be obtained, without contrast, to examine changes in the total volume of the brain as well as the volumes of several brain substructures over time. The MRI may be performed under general anesthesia in this pediatric population. It is important that all procedures requiring general anesthesia are performed in close temporal proximity, while the subject is under anesthesia.
Change from baseline in liver and spleen volume measured using MRI | Baseline through 36 months (3 years)
  If consent if provided, magnetic resonance imaging (MRI) of the abdomen will be obtained, without contrast, to examine changes in the total volume of the liver and spleen over time. The MRI may be performed under general anesthesia in this pediatric population. It is important that all procedures requiring general anesthesia are performed in close temporal proximity, while the subject is under anesthesia.
Change from baseline in liver and spleen volume measured using ultrasound | Baseline through 36 months (3 years)
  Only if consent is not provided to obtain images of the abdomen via MRI, an abdominal ultrasound will be performed to examine changes in the total volume of the liver and spleen over time.

OTHER OUTCOMES:
Exploratory analysis of beta-galactosidase enzyme activity and change over time | Baseline through 36 months (3 years)
  Blood and, if consent is given, cerebrospinal fluid (CSF)* will be collected at the baseline visit and each subsequent visit to analyze beta-galactosidase enzyme activity. The aim is to examine enzyme activity variability, change from baseline and relationship to disease progression. As this biomarker are currently under study, ranges cannot be provided at this time. Additional samples may also be stored at a biobank for future research and testing, if consent is obtained.
  *Collection of CSF via a lumbar puncture is an OPTIONAL procedure conducted only at Baseline and Months 6, 12, 24 and 36.
Exploratory analysis of hexosaminidase enzyme activity and change over time | Baseline through 36 months (3 years)
  Blood and, if consent is given, cerebrospinal fluid (CSF)* will be collected at the baseline visit and each subsequent visit to analyze hexosaminidase enzyme activity. The aim is to examine enzyme activity variability, change from baseline and relationship to disease progression, if applicable. As this biomarker are currently under study, ranges cannot be provided at this time. Additional samples may also be stored at a biobank for future research and testing, if consent is obtained.
  *Collection of CSF via a lumbar puncture is an OPTIONAL procedure conducted only at Baseline and Months 6, 12, 24 and 36.
Exploratory analysis of keratan sulfate levels and change over time | Baseline through 36 months (3 years)
  Blood and urine will be collected at the baseline visit and each subsequent visit to analyze keratan sulfate levels. The aim is to examine variability and change from baseline in the levels as well as relationship to disease progression, if applicable. As this biomarker are currently under study, ranges cannot be provided at this time. Additional samples may also be stored at a biobank for future research and testing, if consent is obtained.
Exploratory analysis of GM1 ganglioside levels and change over time | Baseline through 36 months (3 years)
  If consent is given, cerebrospinal fluid (CSF)* will be collected at the baseline visit and each subsequent visit to analyze GM1 ganglioside levels. The aim is to examine variability and change from baseline in the levels as well as relationship to disease progression. As this biomarker are currently under study, ranges cannot be provided at this time. Additional samples may also be stored at a biobank for future research and testing, if consent is obtained.
  *Collection of CSF via a lumbar puncture is an OPTIONAL procedure conducted only at Baseline and Months 6, 12, 24 and 36.

CONTACTS AND LOCATIONS:
Overall Officials: Can Ficicioglu, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (6):
- United States (2):
  - UCSF Benioff Children's Hospital Oakland, Oakland, California
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Brazil
- Montreal Children's Hospital Research Institute - McGill University, Montreal, Quebec, Canada
- Gazi University, Ankara, Turkey (Türkiye)
- UCL Great Ormond Street Institute of Child Health, London, United Kingdom